CLINICAL TRIAL: NCT05197192
Title: A Prospective, Open-label, Multicentre, Randomized, Phase-3-trial of Acalabrutinib, Obinutuzumab and Venetoclax (GAVE) Compared to Obinutuzumab and Venetoclax (GVE) in Previously Untreated Patients With High Risk Chronic Lymphocytic Leukemia (CLL)
Brief Title: A Phase-3-trial of Acalabrutinib, Obinutuzumab & Venetoclax Compared to Obinutuzumab and Venetoclax in Previously Untreated Patients With High Risk CLL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLL16; 2023-506414-46-00 (EU CTIS Number)
Record Dates: First submitted 2021-09-27; First posted 2022-01-19 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; high risk; tp53 aberration; complex karyotype; unmutated IGHV gene status
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab; venetoclax; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GAVe-Arm (Experimental): Acalabrutinib plus Venetoclax plus Obinutuzumab plus (GAVe)
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax; Drug: Acalabrutinib
- GVe-Arm (Experimental): Obinutuzumab plus Venetoclax (GVe)
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab i.v. infusion:
  Cycle 1 Day 1: Obinutuzumab 100 mg i.v.
  Cycle 1 Day 1 (or 2): Obinutuzumab 900 mg i.v.
  Cycle 1 Day 8: Obinutuzumab 1000 mg i.v.
  Cycle 1 Day 15: Obinutuzumab 1000 mg i.v.
  Cycles 2-6: Day 1: Obinutuzumab 1000 mg i.v.
  Other Names: Gazyva; Gazyvaro
Drug: Venetoclax — Venetoclax p.o.:
  Cycle 1: Days 22-28: Venetoclax 20 mg (2 x 10 mg)
  Cycle 2: Days 1-7: Venetoclax 50 mg (1 x 50 mg)
  Cycle 2:Days 8-14: Venetoclax 100 mg (1 x 100 mg)
  Cycle 2:Days: 15-21: Venetoclax 200 mg (2 x 100 mg)
  Cycle 2:Days: 22-28: Venetoclax 400 mg (4 x 100 mg)
  Cycles 3-12: Days 1-28: Venetoclax 400 mg (4 x 100 mg)
  Other Names: Venclexta; Venclyxto
Drug: Acalabrutinib — Cycles 15-24: Days 1-28:
  100 mg acalabrutinib twice daily p.o. approx. every 12 hrs (corresponding to a total daily dose of 200 mg).
  Other Names: Calquence
  Arms: GAVe-Arm

SUMMARY:
This multicenter, prospective, open-label, randomized, superiority phase 3 study is designed to demonstrate that treatment with a triple combination of acalabrutinib, obinutuzumab and venetoclax (GAVe) prolong the progression-free survival (PFS) as compared to treatment with the combination of obinutuzumab and venetoclax (GVe) in pa-tients with high risk CLL (defined as having at least one of the follow-ing risk factors: 17p-deletion, TP53-mutation, complex karyotype or an unmutated IGHV-gene status).

DETAILED DESCRIPTION:
CLL is the most frequent leukemia in industrialized countries. International guidelines agree on diagnosis and management of this disease. The clinical course of CLL is highly variable and can be predicted by clinical staging (according to Rai and Binet) as well as genetic, serum markers and risk models. This study is designed for a randomized comparison of two different, non-chemotherapeutic and fixed-duration modalities for patients with high risk chronic lymphocytic leukemia (CLL) and addresses a high medical need, since high risk-CLL represents a so far incurable, aggressive cancer. The high risk-group of CLL patients can be identified by molecular characteristics, allowing the inclusion of a clearly described group of patients: 17p-deletion, TP53-mutation and/or complex karyotype.TP53 defects are the strongest prognostic factors for non-response to chemotherapy. Patients harboring TP53 defects should be treated with chemotherapy-free regimens. Complex karyotype (CKT), defined as the presence of three or more chromosomal aberrations in two or more metaphases is associated with a poorer outcome in various hematologic malignancies, including chronic lymphocytic leukemia (CLL). In CLL, CKT is one of several well established adverse prognostic factors, comparable to 17p-deletion, TP53-mutation or unmutated IGHV status. Depending on age and prior exposure to chemotherapy, 10-30% of patients with CLL exhibit CKT. A broad body of evidence has suggested a predictive prognostic value of CKT. Despite considerable advances with chemoimmunotherapy in the treatment of frontline as well as relapsed/refractory (r/r) CLL, outcome of patients with CKT remains poor. To date, a randomized comparison to optimize the treatment of patients with high risk disease defined as either the presence of TP53 aberrations or CKT, by novel agents has not been performed. Patients with high risk CLL (TP53-defects and/or CKT) have a poor outcome with chemoimmunotherapy and do not benefit to the same extent from approved regimen such as continuous treatment of ibrutinib or 12 months treatment with obinutuzumab plus venetoclax. Monotherapy with BTK-inhibitor is less effective in those patients as compared with patients without high risk disease. Venetoclax combined with the anti-CD20 monoclonal antibody obinutuzumab offers a highly effective fixed-duration treatment option with a manageable toxicity profile. The recent results of the CLL14 study define a new standard of a fixed 12-months treatment with obinutuzumab and venetoclax in previously untreated patients yielding a major benefit also for patients with high risk disease as compared to chemoimmunotherapy. However, high risk patients appear to progress earlier than low risk patients and the therapy is not clearly curative so far. Acalabrutinib is a second generation, selective BTK inhibitor which has shown promising overall response rates in patients with relapsed CLL or patients intolerant to ibrutinib. The development of acalabrutinib focussed on minimization of off-target activity. Results of a three-arm study investigating the combination of acalabrutinib plus obinutuzumab versus acalabrutinib alone versus chlorambucil plus obinutuzumab (NCT02475681) showed a substantial improvement of PFS for the combination arm and the monotherapy versus the standard chemoimmunotherapy regimen. The addition of a BTK-inhibitor, such as acalabrutinib to obinutuzumab and venetoclax has the potential to result in a better outcome, because synergistic effects have been reported between BTK inhibitors and B-cell lymphoma 2 (BCL-2) inhibitors or for BCL-2 inhibitors and monoclonal antibodies. Synergistic effects, which are expected to reduce early progressions or insufficient responses, are in particular important for this high risk population. The triple combination of acalabrutinib, obinutuzumab (or rituximab) and venetoclax has been investigated in a phase 1 b- study and had a tolerable safety profile with minimal to no drug-drug interactions, results of a phase 2 trial studying the same combination showed that the triple combination was highly active with 78% undetectable MRD levels in the bone marrow . Currently, the GCLLSG conducts phase 2 studies, investigating a triple combination consisting of BTK- and Bcl2-inhibitors and monoclonal antibodies (CLL2GIVe: NCT02758665; CLL2BAAG: NCT03787264) and a large phase 3 trial with one experimental arm with a triple combination (CLL13, NCT02950051) but results are not yet published. Acalabrutinib, venetoclax and obinutuzumab is now being studied in a registrational phase 3 trial CL-311 (NCT03836261) against the current standard of chemoimmunotherapy (fludarabine/cyclophosphamide/rituximab (FCR), bendamustine/rituximab (BR) in patients without 17p-deletion or TP53-mutation. Acalabrutinib is indicated in Germany as monotherapy or in combination with obinutuzumab for the treatment of adult patients with treatment-naive chronic lymphocytic leukemia (CLL) and as monotherapy for the treatment of adult patients with relapsed chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* Documented CLL/SLL requiring treatment according to iwCLL criteria
* Age at least 18 years
* At least one of the following risk factors: 17p-deletion, TP53-mutation, complex karyotype (defined as defined as the presence of 3 or more chromosomal aberrations in 2 or more metaphases) or an unmutated IGHV gene status.
* Life expectancy ≥ six months
* Adequate bone marrow function indicated by a platelet count >30 x10^9/l
* Creatinine clearance ≥ 30ml/min
* Adequate liver function as indicated by a total bilirubin ≤ 2 x, AST/ ALT ≤ 2.5 x the institutional ULN value, unless directly attributable to the patient's CLL or to Gilbert's Syndrome
* Negative testing for hepatitis B (HbsAg negative and anti-HBc negative; patients positive for anti-HBc may be included if PCR for HBV DNA is negative and HBV-DNA PCR is performed every month until 12 months after last treatment cycle),or hepatitis C (negative testing for hepatitis C RNA within 6 wee
* ks prior to registration for study screening (i.e. PCR only required when serology was positive))
* ECOG (Eastern Cooperative Oncology Group Performance Status) status 0-2

Exclusion Criteria:

* Any prior CLL-specific therapies (except corticosteroid treatment administered due to necessary immediate intervention; within the last 10 days before start of study treatment, only dose equivalents up to 20 mg prednisolone are permitted)
* Absence of high risk disease (17p-deletion, TP53-mutation complex karyotype
* An individual organ/system impairment score of 4 as assessed by the CIRS definition (e.g. advanced cardiac disease (NYHA class 3 or 4) limiting the ability to receive the study treatment or any other life-threatening illness, medical condition or organ system dysfunction that, in the investigator´s opinion, could compromise the patients safety or interfere with the absorption or metabolism of the study drugs (e.g. inability to swallow tablets or impaired resorption in the gastrointestinal tract)
* Transformation of CLL (Richter transformation)
* Malignancies other than CLL currently requiring systemic therapies
* Uncontrolled or active infection of HIV/PML or any other active infection
* Anticoagulant therapy with warfarin or phenoprocoumon
* Pregnant women and nursing mothers

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 50 months after FPI
  The study is designed to demonstrate that 14 cycles of treatment with GAVe followed by up to 10 cycles maintenance with acalabrutinib for patients with detectable MRD at cycle 14 day 14 prolong PFS as compared to 12 cycles of treatment with GVe in patients with high risk CLL (defined as hav-ing at least one of the following risk factors: 17p-deletion, TP53- mutation or complex karyotype).

SECONDARY OUTCOMES:
Minimal residual disease (MRD) levels | 50 months after FPI
  Minimal residual disease (MRD) levels in the peripheral blood (PB) and in the bone marrow (BM) at final restaging ((Staging 5) cycle 15 day 1 for patients in GVe study arm, cycle 14 day 14 for patients in GAVe study arm)
MRD in PB at cycle 27 day 1 | 50 months after FPI
  MRD in PB at cycle 27 day 1 for all patients (end of maintenance for patients in GAVe study arm, who had detectable MRD levels after 14 cycles of GAVe-treatment)
Overall response rate | 50 months after FPI
  Overall response rate (ORR; as per iwCLL guidelines) at cycle 15
Complete response rate | 50 months after FPI
  Complete response rate (CRR; as per iwCLL guidelines) at cycle 15
Overall Survival (OS) | 50 months after FPI
  Overall Survival (OS)
Event-free survival (EFS) | 50 months after FPI
  Event-free survival (EFS)
Duration of response (DOR) | 50 months after FPI
  Duration of response (DOR)
Time to next treatment (TTNT) | 50 months after FPI
  Time to next treatment (TTNT)

OTHER OUTCOMES:
Correlation between MRD in PB/BM and PFS/OS | 50 months after FPI
  Time-to-event analyses will be calculated accordiung to MRD levels in peripheral bloos and bone marrow respectively.
MRD by methods other than flow cytometry (ddPCR) | 50 months after FPI
  New methods of MRD measurements (ddPCR) will be compared with the standard method (flow cytometry )
Correlation between MRD in PB and BM | 50 months after FPI
  MRD levels in the peripheral blood and in the bone marrow will be statistically compared.
Longitudinal Analysis of European Organisation for Research and Treatment of Cancer(EORTC): Quality of Life Questionnaire (QLQ-C30) at defined timepoints | 50 months after FPI
  Outcome measure: scores of EORTC QLQ-C30 and QLQ-CLL17 Questionnaires at defined timepoints will be analyzed and compared to baseline level for each patient. Scoring of the QLQ-C30 is performed according to QLQ-C30 Scoring manual. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Eichhorst, MD, Prof., Principal Investigator — Department I of Internal Medicine, University Hospital Cologne
Locations (30):
- Germany (30):
  - Helios Klinikum Bad Saarow, Bad Saarow
  - DRK Kliniken Berlin Köpenick, Berlin
  - Ev. Diakoniekrankenhaus, Bremen
  - Universitätsklinik Köln, Cologne
  - St. Johannes Hospital, Dortmund
  - Marien Hospital Düsseldorf, Düsseldorf
  - St. Antonius-Hospital, Eschweiler
  - Universitaetsklinikum Essen, Essen
  - Katholisches Krankenhaus Hagen - St. Josefs Hospital, Hagen
  - Universitaetskliniken des Saarlandes, Homburg
  - Klinikum Idar-Oberstein SHG, Idar-Oberstein
  - Staedtisches Klinikum Karlsruhe, Karlsruhe
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Klinikum Landshut, Landshut
  - Klinikum Lippe-Lemgo, Lemgo
  - St Vincenz Krankenhaus, Limburg
  - Universitaetsklinikum Magdeburg, Magdeburg
  - Klinikum Hochsauerland - St. Walburga Krankenhaus, Meschede
  - KH Kliniken Maria Hilf, Mönchengladbach
  - Krankenhaus Muenchen-Schwabing, Munich
  - Klinikum Rechts der Isar - Technische Universitaet Muenchen, Munich
  - Kliniken Ostalb, Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Klinikum Oldenburg, Oldenburg
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Universitätsklinik Rostock, Rostock
  - Caritas-Klinik St. Theresia, Saarbrücken
  - Klinikum Sindelfingen-Böbingen, Sindelfingen
  - Marienhospital Stuttgart, Stuttgart
  - Universitaetsklinik Tuebingen, Tübingen
  - Universitätsklinik Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.dcllsg.com/cll16/